CLINICAL TRIAL: NCT02271191
Title: Effect of Nicardipine on Renal Function in Deliberate Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6-2011-0205
Record Dates: First submitted 2014-10-15; First posted 2014-10-22 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Nicardipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicardipine and Remifentanil (Active Comparator): intravenous nicardipine and remifentanil during deliberate hypotension
  Interventions: Drug: Nicardipine
- Remifentanil (Placebo Comparator): intravenous remifentanil during deliberate hypotension
  Interventions: Drug: Nicardipine

INTERVENTIONS:
Drug: Nicardipine — nicardipine 1-5 ug/kg/min and remifentanil 0.05 ug/kg/min during deliberate hypotension in spine surgery
  Other Names: Perdipine

SUMMARY:
The aim of this study was to demonstrate the effect of nicardipine on renal function with creatinine clearance, serum cystatin C, urine output and fractional excretion of sodium during deliberate hypotension for spine surgery.

DETAILED DESCRIPTION:
To induce deliberate hypotension, pharmacological agents such as inhalation anesthetics, calcium channel blockers, beta-adrenergic blockers have been used alone or in combination. Nicardipine, classed as a calcium channel blocker, has a peripheral vasodilator effect via relaxation of smooth muscle fiber and sympathetic nerve inhibition. Nicardipine expands the renal artery and increases glomerular filtration rate. Previous studies reported the renal protective effect of nicardipine in cardiac surgery with cardiopulmonary bypass and robot-assisted laparoscopic surgery.

The aim of this study was to demonstrate the effect of nicardipine on renal function with creatinine clearance , serum cystatin C, urine output and fractional excretion of sodium during deliberate hypotension for spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing anterior or posterior spine interbody fusion

Exclusion Criteria:

* Patients with American Society of Anesthesiologists physical status III or IV
* Liver dysfunction with aspartate transaminase/alanine transaminase greater than 60/60 IU/L
* Cerebrovascular disease
* Anemia of less than hematocrit 24%
* Diabetes mellitus
* Severe malnutrition
* those diuretics or antihypertensive drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
creatinine clearance | after deliberate hypotension, and POD1
serum cystatin C | before deliberate hypotension, after deliberate hypotension, and POD1
urine output | after deliberate hypotension, and POD1
fractional excretion of sodium | before deliberate hypotension, after deliberate hypotension, and POD1

SECONDARY OUTCOMES:
Risk, injury, failure, loss, and end stage renal disease (RIFLE) criteria | before deliberate hypotension, after deliberate hypotension, and POD1

CONTACTS AND LOCATIONS:
Overall Officials: Chul Ho Chang, MD, PhD, Study Chair — Department of Anesthesiology and Pain Medicine, Gangnam Severance Hospital, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, 211 Eonju-ro, Gangnam-gu, Seoul 135-720, Republic of Korea